CLINICAL TRIAL: NCT02462759
Title: A Phase 2, Randomized, Double-blind, Sham-procedure Controlled Study to Assess the Safety and Tolerability and Explore the Efficacy of ISIS 396443 (BIIB058) Administered Intrathecally in Subjects With Spinal Muscular Atrophy Who Are Not Eligible to Participate in the Clinical Studies ISIS 396443-CS3B or ISIS 396443-CS4
Brief Title: A Study to Assess the Safety and Tolerability of Nusinersen (ISIS 396443) in Participants With Spinal Muscular Atrophy (SMA).
Acronym: EMBRACE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early to roll over participants to open label extension study NCT02594124.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 232SM202; 2014-003657-33 (EudraCT Number)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2015-05-14; First posted 2015-06-04 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: EMBRACE; SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nusinersen (Experimental): Administered by intrathecal injection.
  Interventions: Drug: Nusinersen
- Sham Procedure (Sham Comparator): Small needle prick on the lower back at the location where the IT injection is normally made.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Drug: Nusinersen — Administered by intrathecal injection.
  Other Names: BIIB058; ISIS SMNRx; ISIS 396443; Spinraza
  Arms: Nusinersen
Procedure: Sham Procedure — Small needle prick on the lower back at the location where the IT injection is normally made.
  Arms: Sham Procedure

SUMMARY:
The primary objective of Part 1 of this study is to assess the safety and tolerability of Nusinersen in participants with SMA who are not eligible to participate in the clinical studies ISIS 396443-CS3B (NCT02193074) or ISIS 396443-CS4 (NCT02292537). The secondary objective of Part 1 of this study is to examine the pharmacokinetics (PK) of Nusinersen in participants with SMA. The primary objective of Part 2 of this study is to assess the long-term safety and tolerability of Nusinersen in participants with SMA who participated in Part 1 and completed their End of Part 1 Evaluation assessments. The secondary objective of Part 2 of this study is to examine the PK of Nusinersen in participants with SMA who participated in Part 1 and completed their End of Part 1 Evaluation assessments.

DETAILED DESCRIPTION:
Part 2 is an Open Label extension phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetic documentation of 5q SMA homozygous gene deletion, mutation, or compound heterozygote.
* Onset of clinical signs and symptoms consistent with SMA at ≤6 months of age and have documentation of 3 SMN2 copies OR onset of clinical signs and symptoms consistent with SMA at ≤6 months of age, >7 months of age (211 days) at screening, and have documentation of 2 SMN2 copies OR onset of clinical signs and symptoms consistent with SMA at >6 months of age, are ≤18 months of age at screening, and have documentation of 2 or 3 SMN2 copies.
* Meets age-appropriate institutional criteria for use of anesthesia/sedation, if use is planned for study procedures.
* Medical care, such as routine immunizations meets and is expected to continue to meet guidelines set out in the Consensus Statement for Standard of Care in SMA, in the opinion of the Investigator.
* Participants with 2 SMN2 copies must reside within approximately 9 hours' ground-travel distance from a participating study site for the duration of the study.

Key Exclusion Criteria:

* Meets additional study related criteria.
* Any previous exposure to ISIS 396443; previous dosing in this study or previous studies with ISIS 396443.
* Signs or symptoms of SMA present at birth or within the first week after birth.
* Ventilation for ≥16 hours per day continuously for >21 days at screening.
* Permanent tracheostomy, implanted shunt for CSF drainage, or implanted central nervous system (CNS) catheter at screening.
* History of brain or spinal cord disease that would interfere with the LP procedure, CSF circulation, or safety assessments.
* Hospitalization for surgery (e.g., scoliosis surgery), pulmonary event, or nutritional support within 2 months prior to screening, or hospitalization for surgery planned during the study.
* Clinically significant abnormalities in hematology or clinical chemistry parameters or Electrocardiogram (ECG), as assessed by the Investigator.
* Treatment with an investigational drug for SMA (e.g., albuterol/salbutamol, riluzole, carnitine, sodium phenylbutyrate, valproate, hydroxyurea), biological agent, or device within 30 days prior to screening. Any history of gene therapy, prior antisense oligonucleotide (ASO) treatment, or cell transplantation.

For Part 2 only:

To be eligible to participate in Part 2 of this study, participants must meet the following eligibility criteria at the time of consent to participate in Part 2:

Participation in Part 1 and completion of the End of Part 1 Evaluation assessments.

Ability of parent(s) or legal guardian(s) to understand the purpose and risks of the study and to provide signed and dated informed consent on the Part 2 informed consent form (ICF) and authorization to use confidential health information in accordance with national and local participant privacy regulations.

Able to complete all study procedures, measurements, and visits, and parent or legal guardian/participant has adequately supportive psychosocial circumstances, in the opinion of the Investigator.

Participants will be excluded from the Part 2 if they meet the following exclusion criterion at the time of consent into Part 2 of the study:

Any significant change in clinical status, including laboratory tests that, in the opinion of the Investigator, would make them unsuitable to participate in Part 2. The Investigator must reassess the subject's medical fitness for participation and consider any diseases that would preclude treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (7):
- United States (6):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Connecticut Childrens Medical, Hartford, Connecticut
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Research Institute, Seattle, Washington
- LMU-Campus Innenstadt, München, Germany

REFERENCES:
- [Derived] Acsadi G, Crawford TO, Muller-Felber W, Shieh PB, Richardson R, Natarajan N, Castro D, Ramirez-Schrempp D, Gambino G, Sun P, Farwell W. Safety and efficacy of nusinersen in spinal muscular atrophy: The EMBRACE study. Muscle Nerve. 2021 May;63(5):668-677. doi: 10.1002/mus.27187. Epub 2021 Feb 16. PMID 33501671
- See also: Clinical Study Report (CSR) Synopsis - a results summary — http://clinicalresearch.biogen.com/Content/Studies/232SM202%20Biogen.comPacket_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from sites in the US and Germany. Part 1 was terminated early as positive efficacy results were observed in interim analysis of study NCT02193074 and it was considered unethical to continue this part of study. Part 2 was also terminated early to rollover and continue to follow participants in study NCT02594124.
Pre-assignment Details: Total of 21 participants with SMA were randomized in Part 1 of the study(7 participants in sham procedure group,14 participants in ISIS 396443 group).1 participant died in sham procedure group of Part 1.Total of 20 participants were enrolled to receive ISIS 396443 in open-label phase of Part 2.Integrated analysis was performed for Part 1 and 2.
Groups:
- Sham Procedure (Part 1): Sham procedure on Day 1, 15, 29, 64, 183 and 302.
- ISIS 396443 (Part 1): Single dose of 9.6 milligrams (mg) to 12.0 mg ISIS 396443, based on participant's age, intrathecal bolus injection loading doses on Day 1, 15, 29, 64 and maintenance doses, every 4 months, on Day 183 and 302.
- ISIS 396443 (Part 2): Participants who were in Sham procedure group in Part 1, received single dose of 12.0 mg ISIS 396443 intrathecal bolus injection loading doses on Day 1, 15, 29, 64 and maintenance doses, every 4 months, on Day 183, 302, 421, 540, 659 and 778 in Part 2; participants who were in ISIS 396443 group in Part 1 continued to receive a single dose of 9.6 mg to 12.0 mg ISIS 396443 intrathecal bolus injection maintenance doses on Day 1, 120, 239, 358, 477, 596 and 715 in Part 2.
Period: Part 1: Double Blind
Arm/Group | Sham Procedure (Part 1) | ISIS 396443 (Part 1) | ISIS 396443 (Part 2)
Started | 7 | 14 | 0
Completed | 6 | 14 | 0
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Period: Part 2: Open-Label Phase
Arm/Group | Sham Procedure (Part 1) | ISIS 396443 (Part 1) | ISIS 396443 (Part 2)
Started | 0 | 0 | 20
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population include all participants who were randomized, receive at least 1 dose of ISIS 396443 or sham procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Procedure (Part 1) | ISIS 396443 (Part 1) | Total
Number analyzed (Participants) | 7 | 14 | 21
Age, Continuous [Mean (Standard Deviation); unit: months] | 24.4 (13.83) | 19.4 (10.12) | 21.1 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 2 | 9 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 2 | 1 | 3
  Ethnicity: Not Hispanic or Latino | 4 | 9 | 13
  Ethnicity: Not reported due to confidentiality | 1 | 4 | 5
  Race: Asian | 3 | 2 | 5
  Race: White | 2 | 7 | 9
  Race: Other | 1 | 1 | 2
  Race: Not reported due to confidentiality | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A SAE is any untoward medical occurrence that at any dose results in death, life-threatening event, requires inpatient hospitalization, significant disability/incapacity or congenital anomaly.
Time Frame: Part 1 and 2: From first dose/sham procedure to end of study (up to 1080 days)
Population: The safety population included all participants who were randomized and received at least 1 dose of study treatment or sham procedure.
Measure: Count of Participants; unit: Participants
Groups:
- Sham Procedure in Part 1: Participants who received single dose of sham procedure on Day 1, 15, 29, 64, 183 and 302 in Part 1 of the study.
- ISIS 396443 Part 2(Participants on Sham in Part 1): Participants who received single dose of ISIS 396443 on Day 1, 15, 29, 64, 183, 302, 421, 540, 659 and 778 in Part 2.
- ISIS 396443 Part 1 & 2: Participants who received single dose of ISIS 396443 on Day 1, 15, 29, 64, 183 and 302 in Part 1 of the study and then received single dose of ISIS 396443 on Day 1, 120, 239, 358, 477, 596 and 715 in Part 2 of the study.
Arm/Group | Sham Procedure in Part 1 | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 7 | 6 | 14
Participants
  AEs | 6 | 6 | 14
  SAEs | 3 | 4 | 9

2. Primary Outcome: Number of Participants With Change From Baseline in Clinical Laboratory Parameters
Description: Clinically significant changes in laboratory parameters were evaluated for assessing the safety of ISIS 396443.
Time Frame: Part 1 and 2: From first dose/sham procedure to end of study (up to 1080 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Procedure in Part 1 | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 7 | 6 | 14
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Change From Baseline in Electrocardiograms (ECGs)
Description: Clinically significant changes in ECG measurements were evaluated for assessing the safety of ISIS 396443.
Time Frame: Part 1: Day 2, 29 and 422; Part 2: Day 1 to 596
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Procedure in Part 1 | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 7 | 6 | 14
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Change From Baseline in Vital Signs
Description: Clinically significant changes in vital signs were evaluated for assessing the safety of ISIS 396443. Vital signs that were assessed included resting systolic and diastolic blood pressure, pulse rate, respiratory rate, temperature, pulse oximetry, and transcutaneous carbon dioxide.
Time Frame: Part 1: Day 2, 29 and 422; Part 2: Day 1 to 596
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Procedure in Part 1 | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 7 | 6 | 14
Participants | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Head Circumference
Description: Participants were analyzed for change in growth parameter of head circumference to evaluate clinical efficacy. WHO Child Growth Standards were used to determine the head circumference percentile. Study days were windowed for integrated analysis and labelled as follows: Days <=1 as Baseline; Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Part 2: Baseline, Day 15, 29, 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: Safety population: participants who were randomized and received at least 1 dose of study treatment or sham procedure. Number analyzed indicates participants who were evaluated for the specified time points. Due the early termination of Part 2, no participants in the ISIS 396443 Part 2(participants on sham in Part 1) were on study beyond Day 659.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
centimeter (cm)
  Baseline | 50.8 (3.83) | 47.3 (1.51)
  Change at Day 15: number analyzed (Participants) | 5 | 14
  Change at Day 15 | -0.7 (3.34) | 0.1 (0.36)
  Change at Day 29: number analyzed (Participants) | 6 | 13
  Change at Day 29 | 0.0 (2.76) | 0.3 (0.65)
  Change at Day 64 | 0.1 (2.64) | 0.5 (0.73)
  Change at Day 183 | 0.3 (3.10) | 1.0 (1.12)
  Change at Day 302 | 1.0 (3.28) | 1.6 (1.05)
  Change at Day 422: number analyzed (Participants) | 6 | 13
  Change at Day 422 | 0.9 (2.47) | 2.0 (1.24)
  Change at Day 540 | 1.3 (1.97) | 2.5 (1.24)
  Change at Day 659 | 1.5 (2.53) | 2.6 (1.37)
  Change at Day 778: number analyzed (Participants) | 0 | 14
  Change at Day 778 |  | 2.8 (0.92)
  Change at Day 898: number analyzed (Participants) | 0 | 12
  Change at Day 898 |  | 3.5 (1.05)
  Change at Day 1018: number analyzed (Participants) | 0 | 5
  Change at Day 1018 |  | 3.5 (2.06)
  Change at Day 1138: number analyzed (Participants) | 0 | 1
  Change at Day 1138 |  | 4.0 (0)

6. Primary Outcome: Change From Baseline in Chest Circumference
Description: Participants were analyzed for change in growth parameter of chest circumference to evaluate clinical efficacy. WHO Child Growth Standards were used to determine the chest circumference percentile. Study days were windowed for integrated analysis and labelled as follows: Days <=1 as Baseline; Days>1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Part 2: Baseline, Day 15, 29, 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
cm
  Baseline | 51.3 (5.45) | 46.9 (3.91)
  Change at Day 15: number analyzed (Participants) | 5 | 14
  Change at Day 15 | -0.2 (3.86) | -0.4 (1.53)
  Change at Day 29: number analyzed (Participants) | 6 | 13
  Change at Day 29 | -1.1 (2.70) | 0.2 (1.39)
  Change at Day 64 | -0.9 (3.50) | 0.2 (1.92)
  Change at Day 183 | 0.2 (3.04) | 1.4 (2.02)
  Change at Day 302 | 1.2 (3.07) | 1.6 (2.86)
  Change at Day 422 | 0.5 (3.72) | 2.8 (2.73)
  Change at Day 540 | 1.8 (2.42) | 3.8 (3.23)
  Change at Day 659 | 2.9 (3.85) | 5.1 (3.29)
  Change at Day 778: number analyzed (Participants) | 0 | 14
  Change at Day 778 |  | 5.5 (3.52)
  Change at Day 898: number analyzed (Participants) | 0 | 12
  Change at Day 898 |  | 7.1 (3.04)
  Change at Day 1018: number analyzed (Participants) | 0 | 5
  Change at Day 1018 |  | 9.7 (4.92)
  Change at Day 1138: number analyzed (Participants) | 0 | 1
  Change at Day 1138 |  | 9.1 (0)

7. Primary Outcome: Change From Baseline in Arm Circumference
Description: Participants were analyzed for change in growth parameter of arm circumference to evaluate clinical efficacy. WHO Child Growth Standards were used to determine the arm circumference percentile. Study days were windowed for integrated analysis and labelled as follows: Days <=1 as Baseline; Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Part 2: Baseline, Day 15, 29, 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
cm
  Baseline | 16.2 (1.19) | 14.5 (1.85)
  Change at Day 15: number analyzed (Participants) | 5 | 14
  Change at Day 15 | -0.4 (1.04) | 0.3 (0.61)
  Change at Day 29: number analyzed (Participants) | 6 | 13
  Change at Day 29 | -0.5 (1.08) | -0.1 (0.54)
  Change at Day 64 | -0.3 (0.49) | -0.4 (0.89)
  Change at Day 183 | 0.0 (0.89) | 0.0 (0.85)
  Change at Day 302 | -0.6 (0.89) | 0.2 (1.17)
  Change at Day 422 | -0.6 (1.82) | 0.5 (1.71)
  Change at Day 540 | -0.2 (2.24) | 0.5 (1.89)
  Change at Day 659 | 0.6 (0.93) | 0.6 (1.93)
  Change at Day 778: number analyzed (Participants) | 0 | 14
  Change at Day 778 |  | 0.0 (2.18)
  Change at Day 898: number analyzed (Participants) | 0 | 12
  Change at Day 898 |  | 0.8 (2.70)
  Change at Day 1018: number analyzed (Participants) | 0 | 5
  Change at Day 1018 |  | 1.0 (2.02)
  Change at Day 1138: number analyzed (Participants) | 0 | 1
  Change at Day 1138 |  | 1.5 (0)

8. Primary Outcome: Change From Baseline in Weight for Age
Description: Participants were analyzed for change in growth parameter of weight for age to evaluate clinical efficacy. WHO Child Growth Standards were used to determine the weight for age percentile. Study days were windowed for integrated analysis and labelled as follows: Days <=1 as Baseline; Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Part 2: Baseline, Day 15, 29, 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
kilogram (kg)
  Baseline | 42.5 (40.87) | 25.3 (28.41)
  Change at Day 15 | -1.3 (1.41) | 3.6 (12.12)
  Change at Day 29 | -2.4 (1.61) | -1.4 (4.82)
  Change at Day 64 | -2.9 (2.58) | 0.5 (8.17)
  Change at Day 183 | -3.8 (6.93) | -5.9 (8.73)
  Change at Day 302 | -10.1 (13.04) | -8.0 (15.42)
  Change at Day 422 | -6.3 (9.45) | -7.5 (17.52)
  Change at Day 540 | -7.0 (6.56) | -8.1 (17.26)
  Change at Day 659 | -8.5 (17.64) | -10.5 (22.23)
  Change at Day 778: number analyzed (Participants) | 0 | 14
  Change at Day 778 |  | -13.2 (16.95)
  Change at Day 898: number analyzed (Participants) | 0 | 12
  Change at Day 898 |  | -10.5 (24.10)
  Change at Day 1018: number analyzed (Participants) | 0 | 5
  Change at Day 1018 |  | -7.0 (34.14)
  Change at Day 1138: number analyzed (Participants) | 0 | 1
  Change at Day 1138 |  | 0.3 (0)

9. Primary Outcome: Change From Baseline in Weight
Description: Participants were analyzed for change in growth parameter of weight to evaluate clinical efficacy. WHO Child Growth Standards were used to determine the weight percentile. Study days were windowed for integrated analysis and labelled as follows: Days <=1 as Baseline; Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Part 2: Baseline, Day 15, 29, 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
kg
  Baseline | 13.0 (2.00) | 9.5 (1.37)
  Change at Day 15 | -0.1 (0.23) | 0.2 (0.44)
  Change at Day 29 | -0.1 (0.26) | 0.1 (0.23)
  Change at Day 64 | 0.0 (0.39) | 0.4 (0.42)
  Change at Day 183 | 0.8 (0.61) | 0.7 (0.48)
  Change at Day 302 | 0.7 (1.04) | 1.3 (0.87)
  Change at Day 422 | 1.8 (1.03) | 1.9 (1.02)
  Change at Day 540 | 2.3 (1.33) | 2.2 (1.17)
  Change at Day 659 | 3.1 (1.39) | 2.8 (1.41)
  Change at Day 778: number analyzed (Participants) | 0 | 14
  Change at Day 778 |  | 3.2 (1.87)
  Change at Day 898: number analyzed (Participants) | 0 | 12
  Change at Day 898 |  | 3.9 (2.86)
  Change at Day 1018: number analyzed (Participants) | 0 | 5
  Change at Day 1018 |  | 4.3 (1.96)
  Change at Day 1138: number analyzed (Participants) | 0 | 1
  Change at Day 1138 |  | 5.0 (0)

10. Primary Outcome: Change From Baseline in Head to Chest Circumference (HCC) Ratio
Description: Participants were analyzed for change in growth parameter of HCC to evaluate clinical efficacy. WHO Child Growth Standards were used to determine the HCC circumference percentile. Study days were windowed for integrated analysis and labelled as follows: Days <=1 as Baseline; Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Part 2: Baseline, Day 15, 29, 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
ratio
  Baseline | 1.0 (0.05) | 1.0 (0.08)
  Change at Day 15: number analyzed (Participants) | 5 | 14
  Change at Day 15 | 0.0 (0.03) | 0.0 (0.03)
  Change at Day 29: number analyzed (Participants) | 6 | 13
  Change at Day 29 | 0.0 (0.04) | 0.0 (0.04)
  Change at Day 64 | 0.0 (0.04) | 0.0 (0.05)
  Change at Day 183 | 0.0 (0.05) | 0.0 (0.05)
  Change at Day 302 | 0.0 (0.03) | 0.0 (0.06)
  Change at Day 422: number analyzed (Participants) | 6 | 13
  Change at Day 422 | 0.0 (0.04) | 0.0 (0.06)
  Change at Day 540 | 0.0 (0.03) | 0.0 (0.06)
  Change at Day 659 | 0.0 (0.03) | -0.1 (0.06)
  Change at Day 778: number analyzed (Participants) | 0 | 14
  Change at Day 778 |  | -0.1 (0.07)
  Change at Day 898: number analyzed (Participants) | 0 | 12
  Change at Day 898 |  | -0.1 (0.06)
  Change at Day 1018: number analyzed (Participants) | 0 | 5
  Change at Day 1018 |  | -0.1 (0.10)
  Change at Day 1138: number analyzed (Participants) | 0 | 1
  Change at Day 1138 |  | -0.1 (0)

11. Primary Outcome: Change From Baseline in Body Length
Description: Participants were analyzed for change in growth parameter of body length to evaluate clinical efficacy. WHO Child Growth Standards were used to determine the body length percentile. Study days were windowed for integrated analysis and labelled as follows: Days <=1 as Baseline; Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Part 2: Baseline, Day 15, 29, 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
cm
  Baseline | 95.0 (9.48) | 79.9 (5.25)
  Change at Day 15: number analyzed (Participants) | 5 | 14
  Change at Day 15 | -1.6 (3.19) | -0.1 (1.81)
  Change at Day 29: number analyzed (Participants) | 6 | 13
  Change at Day 29 | -0.9 (3.49) | 0.9 (1.66)
  Change at Day 64 | 0.5 (4.77) | 1.8 (2.40)
  Change at Day 183 | 3.0 (4.16) | 5.6 (2.36)
  Change at Day 302 | 2.9 (5.76) | 7.1 (2.70)
  Change at Day 422 | 4.2 (5.42) | 9.3 (3.09)
  Change at Day 540 | 4.6 (7.18) | 11.6 (3.93)
  Change at Day 659 | 10.8 (4.12) | 13.1 (3.79)
  Change at Day 778: number analyzed (Participants) | 0 | 14
  Change at Day 778 |  | 14.8 (3.94)
  Change at Day 898: number analyzed (Participants) | 0 | 12
  Change at Day 898 |  | 17.2 (5.62)
  Change at Day 1018: number analyzed (Participants) | 0 | 5
  Change at Day 1018 |  | 19.0 (6.67)
  Change at Day 1138: number analyzed (Participants) | 0 | 1
  Change at Day 1138 |  | 15.8 (0)

12. Primary Outcome: Number of Participants With Change From Baseline in Neurological Examination Outcomes
Description: Neurological examinations included assessment of mental status, level of consciousness, sensory function, motor function, cranial nerve function, reflexes, mood, speech/language and hearing.
Time Frame: Part 1: Baseline to Day 422; Part 2: Baseline to Day 596
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Procedure in Part 1 | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 7 | 6 | 14
Participants
  Mental Status | 0 | 1 | 3
  Level of consciousness | 0 | 1 | 2
  Sensory function | 0 | 0 | 0
  Motor function | 0 | 0 | 0
  Cranial nerve function: Eye Movement | 0 | 0 | 1
  Cranial nerve function: Vision | 0 | 0 | 1
  Reflexes | 0 | 0 | 0
  Mood | 5 | 5 | 12
  Speech/Language | 0 | 1 | 1
  Hearing | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Change From Baseline in Activated Partial Thromboplastin Time [aPTT]
Description: Activated partial thromboplastin time was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of aPTT at baseline to low values postbaseline. "Shift to high" measured change in normal, high and unknown values of aPTT at baseline to high values postbaseline.
Time Frame: Part 2: Up to 1080 days
Population: The safety population included all participants who were randomized and received at least 1 dose of study treatment or sham procedure. Number analyzed indicates participants whose baseline value was not low (or high) and who had at least one post-baseline measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
Participants
  Shift to Low: number analyzed (Participants) | 6 | 9
  Shift to Low | 0 | 0
  Shift to High: number analyzed (Participants) | 6 | 10
  Shift to High | 0 | 0

14. Primary Outcome: Number of Participants With Change From Baseline in Partial Thromboplastin Time [PTT]
Description: PTT was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of PTT at baseline to low values postbaseline. "Shift to high" measured change in normal, high and unknown values of PTT at baseline to high values postbaseline.
Time Frame: Part 2: Up to 1080 days
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
Participants
  Shift to Low: number analyzed (Participants) | 5 | 6
  Shift to Low | 0 | 0
  Shift to High: number analyzed (Participants) | 5 | 6
  Shift to High | 0 | 0

15. Primary Outcome: Number of Participants With Change From Baseline in International Normalized Ratio [INR])
Description: INR was evaluated to assess safety. "Shift to low" measured change in normal, high and unknown values of INR at baseline to low values postbaseline. "Shift to high" measured change in normal, high and unknown values of INR at baseline to high values postbaseline.
Time Frame: Part 2: Up to 1080 days
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
Participants
  Shift to Low: number analyzed (Participants) | 4 | 7
  Shift to Low | 0 | 0
  Shift to High: number analyzed (Participants) | 4 | 7
  Shift to High | 0 | 0

16. Primary Outcome: Number of Participants With Presence of Urine Total Protein Post-baseline
Description: Urine total protein was evaluated to assess safety.
Time Frame: Part 2: Up to 1080 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
Participants
  Baseline | 0 | 1
  High/Postive | 2 | 8

17. Secondary Outcome: Plasma Concentration of ISIS 396443 in Part 2 of Study in Participants Who Received Sham Procedure in Part 1 of the Study
Description: Study days were windowed for integrated analysis and labelled as follows: Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659.
Time Frame: Pre-dose on Days 64, 183, 540 and 659
Population: The pharmacokinetic (PK) population included all participants who were randomized and have at least 1 evaluable post dose or post sham-procedure PK sample.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1)
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL)
  Day 64 | 1.983 (0.7320)
  Day 183 | 0.776 (0.3994)
  Day 540 | 0.425 (0.2200)
  Day 659 | 0.365 (0.1146)

18. Secondary Outcome: Plasma Concentration of ISIS 396443 in Part 1 and 2 of Study in Participants Who Received ISIS 396443 in Part 1 of the Study
Description: Study days were windowed for integrated analysis and labelled as follows: Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018;Days >1078 to <= 1198 as Day 1138.
Time Frame: Pre-dose on Days 64, 183, 302, 422, 540, 659, 778, 898, 1018 and 1138
Population: The PK population included all participants who were randomized and have at least 1 evaluable post dose or post sham-procedure PK sample. Number analyzed indicates participants who were evaluated for the specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 14
ng/mL
  Day 64 | 2.139 (0.8811)
  Day 183: number analyzed (Participants) | 13
  Day 183 | 1.059 (0.5569)
  Day 302: number analyzed (Participants) | 5
  Day 302 | 0.667 (0.1852)
  Day 422: number analyzed (Participants) | 9
  Day 422 | 0.858 (0.4636)
  Day 540: number analyzed (Participants) | 5
  Day 540 | 0.608 (0.2736)
  Day 659: number analyzed (Participants) | 9
  Day 659 | 0.739 (0.2812)
  Day 778: number analyzed (Participants) | 5
  Day 778 | 0.590 (0.3414)
  Day 898: number analyzed (Participants) | 10
  Day 898 | 0.661 (0.2558)
  Day 1018: number analyzed (Participants) | 4
  Day 1018 | 0.329 (0.1020)
  Day 1138: number analyzed (Participants) | 1
  Day 1138 | 0.423 (0)

19. Secondary Outcome: Cerebrospinal Fluid (CSF) Concentration of ISIS 396443 in Part 2 of Study in Participants Who Received Sham Procedure in Part 1 of the Study
Description: CSF samples were analyzed for ISIS 396443 concentrations in participants. Study days were windowed for integrated analysis and labelled as follows: Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540.
Time Frame: Pre-dose on Days 15, 29, 64, 183, 302, 422 and 540
Population: as for outcome 18
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1)
Number analyzed (Participants) | 6
ng/mL
  Day 1: number analyzed (Participants) | 5
  Day 1 | NA (NA) — Mean was below the lower limit of quantification (LLOQ) hence standard deviation was not evaluated. LLOQ is 50 picogram per millilitre.
  Day 15: number analyzed (Participants) | 5
  Day 15 | 3.094 (1.2172)
  Day 29 | 4.805 (2.6706)
  Day 64 | 4.357 (2.3229)
  Day 183 | 4.110 (2.4535)
  Day 302 | 5.397 (2.7503)
  Day 422 | 6.460 (2.9428)
  Day 540 | 8.405 (6.2423)

20. Secondary Outcome: CSF Concentration of ISIS 396443 in Part 1 and 2 of Study in Participants Who Received ISIS 396443 in Part 1 of the Study
Description: CSF samples were analyzed for ISIS 396443 concentrations in participants. Study days were windowed for integrated analysis and labelled as follows: Days >1 to <= 22 as Day 15;Days >22 to <=47 as Day 29;Days >47 to <= 123 as Day 64;Days >123 to <=242 as Day 183;Days >242 to <=362 as Day 302;Days >362 to <=482 as Day 422;Days >482 to <= 600 as Day 540;Days >600 to <= 719 as Day 659;Days >719 to <= 838 as Day 778;Days >838 to <= 958 as Day 898;Days >958 to <= 1078 as Day 1018.
Time Frame: Pre-dose on Days 15, 29, 64, 183, 302, 422, 540, 659, 778, 898 and 1018
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 14
ng/mL
  Day 1: number analyzed (Participants) | 8
  Day 1 | NA (NA) — Mean was below the lower limit of quantification (LLOQ) hence standard deviation was not evaluated. LLOQ is 50 picogram per millilitre.
  Day 15: number analyzed (Participants) | 13
  Day 15 | 3.925 (2.0525)
  Day 29 | 7.273 (4.4786)
  Day 64 | 7.176 (2.8487)
  Day 183 | 8.226 (3.6450)
  Day 302: number analyzed (Participants) | 13
  Day 302 | 8.968 (3.1188)
  Day 422: number analyzed (Participants) | 13
  Day 422 | 9.251 (4.0631)
  Day 540 | 9.026 (2.6864)
  Day 659 | 9.785 (3.3725)
  Day 778: number analyzed (Participants) | 13
  Day 778 | 8.632 (2.4131)
  Day 898: number analyzed (Participants) | 8
  Day 898 | 11.321 (8.9351)
  Day 1018: number analyzed (Participants) | 1
  Day 1018 | 7.010 (0)

21. Secondary Outcome: Number of Participants With Plasma Antibodies to ISIS 396443
Time Frame: Part 2: Baseline to Day 596
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ISIS 396443 Part 2(Participants on Sham in Part 1) | ISIS 396443 Part 1 & 2
Number analyzed (Participants) | 6 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From start to end of study (up to 1133 days)
Description: The safety population included all participants who were randomized and received at least 1 dose of study treatment or sham procedure.
Arm/Group | Sham Procedure in Part 1 | ISIS 396443 Part 1 & 2 | ISIS 396443 Part 2(Participants on Sham in Part 1)
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/7 | 9/14 | 4/6
Other Adverse Events (participants affected / at risk) | 6/7 | 14/14 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Procedure in Part 1 (N=7) | ISIS 396443 Part 1 & 2 (N=14) | ISIS 396443 Part 2(Participants on Sham in Part 1) (N=6)
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Brain death (General disorders) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Bronchitis moraxella (Infections and infestations) | 0 | 0 | 1
Enterovirus infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 7 | 3
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 1
Pneumonia moraxella (Infections and infestations) | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 2 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Rhinovirus infection (Infections and infestations) | 1 | 2 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Procedure in Part 1 (N=7) | ISIS 396443 Part 1 & 2 (N=14) | ISIS 396443 Part 2(Participants on Sham in Part 1) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 3 | 0
Congenital nystagmus (Congenital, familial and genetic disorders) | 0 | 1 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Myopia (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0
Oral contusion (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 1
Teething (Gastrointestinal disorders) | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 7 | 2
Asthenia (General disorders) | 0 | 2 | 0
Complication associated with device (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 12 | 4
Swelling (General disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 4 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 5 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 5 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 2 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 7 | 2
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1
Pneumonia moraxella (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 3 | 1
Respiratory tract infection (Infections and infestations) | 1 | 5 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 9 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 5 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 3 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspiration bronchial (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0
Bone density decreased (Investigations) | 0 | 0 | 1
Carnitine decreased (Investigations) | 0 | 1 | 0
Enterobacter test positive (Investigations) | 0 | 1 | 0
Full blood count increased (Investigations) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 2 | 0
Oxygen saturation decreased (Investigations) | 0 | 2 | 1
Pco2 increased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0
Urine output increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1
Weight increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 0
Device extrusion (Product Issues) | 0 | 1 | 0
Dysphemia (Psychiatric disorders) | 0 | 0 | 1
Intermittent explosive disorder (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Penile adhesion (Reproductive system and breast disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Despite the early termination of both Parts of the study, the data from this study is of quality and reliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT02462759/SAP_000.pdf
  • Study Protocol (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT02462759/Prot_001.pdf